CLINICAL TRIAL: NCT00495040
Title: Phase II Escalated/Accelerated Proton Radiotherapy for Inoperable Stage I (T1-T2, N0, M0) and Selected Stage II (T3N0M0) Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Proton Radiotherapy for Patients With Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0977; NCI-2012-01503 (Registry Identifier: NCI CTRP); P01CA021239-30 (NIH)
Record Dates: First submitted 2007-06-28; First posted 2007-07-02 (Estimated); Results first posted 2019-01-14 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2018-12

CONDITIONS: Lung Cancer
Keywords: Non-Small Cell Lung Cancer; Lung Cancer; Proton Radiotherapy; Proton Beam; NSCLC
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Proton Radiotherapy (Experimental): Proton radiotherapy 87.5 CGE with 2.5 Gy/fraction for 35 treatments.
  Interventions: Radiation: Proton Radiotherapy

INTERVENTIONS:
Radiation: Proton Radiotherapy — 87.5 CGE with 2.5 Gy/fraction for 35 treatments

SUMMARY:
The goal of this clinical research study is to learn if escalated/accelerated proton radiotherapy can improve the control of Non-Small Cell Lung Cancer (NSCLC) and decrease side effects. The safety of this treatment will also be studied.

Objectives:

To assess the therapeutic efficacy and toxicities of proton radiotherapy with escalated/accelerated dose for patients with medically inoperable stage I (T1-2, N0,M0) NSCLC.

Primary goals:

1. Improve 2 years progression free survival at the primary site, and
2. reduce acute and chronic toxicity

Secondary goals:

1. Improve disease specific survival at 2 years.
2. Study the potential of pre- and post treatment PET/CT in predicting clinical outcome.
3. Study the role of biomarkers in predicting therapeutic response and toxicities.

DETAILED DESCRIPTION:
A proton beam is made up of charged particles that have a well-defined range of penetration into tissues. How deep it can penetrate is decided by both the beam's energy and the density of the tissue through which it passes. As the proton beam penetrates the body, the particles slow down, and the beam deposits its dose sharply near the end of its range. This is a phenomenon known as the Bragg peak. By adjusting the Bragg peak, the doctor can deliver a full, localized, uniform dose of energy to the treatment site while sparing the surrounding normal tissues. The proton beam is ideal for treatments where organ preservation is very important, such as lung cancer. Researchers know that standard photon radiotherapy is not able to adequately control tumor growth. But unfortunately, it is not possible to increase the dose of photon radiotherapy without also significantly increasing the side effects. In this study, using proton radiotherapy, researchers will increase the dose about 40% higher than standard photon radiotherapy.

Screening Tests

Signing this consent form does not mean that you will be able to take part in this study. You will have "screening tests" to help the doctor decide if you are eligible to take part in this study. The following tests and procedures will be performed before starting treatment on this study:

Your complete medical history will be recorded. You will have a physical exam. Blood (about 4 teaspoons) will be drawn (within 30 days) for the routine blood tests You will have a computed tomography (CT) scan or positron emission tomography (PET/CT) scan of the chest, an MRI scan or CT of the brain, You will have a lung function test. Women who are able to have children must have a negative blood-pregnancy test. You will have a 4DCT.

Study Drug Administration If you are found to be eligible to take part in this study, you will receive 35 treatments of proton radiotherapy (radiotherapy does not have to start on a Monday but it cannot start on a Friday; usually Monday through Thursday for 7 to 8 weeks). During the treatment, you will lie still on a table for about 30-45 minutes per day in the same position. The proton machine will deliver the dose according to the plan designed by the physician and controlled by a computer. You will not feel, see, or smell anything during the proton beam delivery.

During the treatment, you will be seen by a doctor and research nurse once a week to evaluate possible side effects. You will have a physical exam and you will have a medical history.

You will be taken off study early if the disease gets worse or intolerable side effects occur. After finishing the treatment, follow up is recommended 6 weeks after completion of radiotherapy, required every 3 months (+/-1 month) for two years, then every (+/-1 month) 6 months for three years, and then once a year for 2 years. You will have imaging tests (chest CT or PET scan), lung function test and routine blood tests (about 2 teaspoons) at the follow-up visits. You are allowed to have further chemotherapy or other treatment while you are still in the follow-up on this study. You should discuss chemotherapy with your medical oncologist.

This is an investigational study. Proton radiotherapy is FDA approved for the treatment of lung cancer treatment. Up to 40 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically documented NSCLC.
2. Patients with inoperable centrally located tumors, defined as those within 2 cm of the bronchial tree, major vessels, esophagus, heart, or other mediastinal structures but no direct invasion, T1N0M0 (stage IA), or any location of T2N0M0 (stage IB) and T3N0M0 (selected stage II with chest wall involvement) NSCLC.
3. Performance score KPS 60-100.

Exclusion Criteria:

1. Prior radiotherapy to the chest.
2. Previous or concomitant malignancy other than (a) curatively treated carcinoma in situ of cervix, (b) basal cell carcinoma of the skin, (c) curatively treated superficial transitional cell carcinoma of the urinary bladder, and (d) early stage tumor treated more than 3 years ago for cure.
3. Pregnancy. Patients, both men and women of child bearing potential should use an effective method of birth control throughout their participation in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2006-05-04 (Actual); Primary Completion 2017-06-14 (Actual); Study Completion 2017-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joe Y. Chang, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: (1)Inoperable NSCLC;(2)T1N0M0 (stage IA) that was centrally or superiorly located ≤ 2 cm in all directions of any critical mediastinal structure; T2N0M0 in any location (stage IB, tumor size>3 cm, with no upper size limit), or selected T3N0M0 (stage II,chest wall, mediastinal pleura, or parietal pericardium involvement) in any location (3)ECOG≤2
Groups:
- Dose-escalated Proton Therapy for Early-stage NSCLC: 35 patients were treated with 87.5 Gy at 2.5 Gy/fraction of proton therapy, with fraction given once a day, 5 days per week. The biological effective dose was 109.4 Gy using α/β of 10
Period: Overall Study
Arm/Group | Dose-escalated Proton Therapy for Early-stage NSCLC
Started | 38
Completed | 35
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: There were 35 out of 38 patients treated under the protocol and evaluable for data analysis.
Groups:
- Dose-escalated Proton Therapy for Early-stage Non-small Cell l: 35 patients were treated with 87.5 Gy at 2.5 Gy/fraction of proton therapy, with fraction given once a day, 5 days per week. The biological effective dose was 109.4 Gy using α/β of 10
Arm/Group | Dose-escalated Proton Therapy for Early-stage Non-small Cell l
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 35
Age [Median (Full Range); unit: years] — Population: There were 35 out of 38 patients treated under the protocol and evaluable for data analysis.
  years | 73 [66 to 83]
Karnofsky Performance Status (KPS) Score [Median (Full Range); unit: units on a scale (%)] — This is phase I/II one arm study. The focus is safety and tolerability (toxicity). Therefore, there are no results about factors and better or worse outcome. Population: The Karnofsky Performance Score (KPS) ranking runs from 100 to 0, where 100 is "perfect" Normal health and 0 is death. Practitioners occasionally assign performance scores in between standard intervals of 10. The KPS was to allow physicians to evaluate a patient's survival. The higher KPS scores, the better treatment outcome.
  units on a scale (%) | 80 [60 to 90]
Gross Tumor Volume (GTV) [Median (Full Range); unit: cubic centimeters] — This is phase I/II one arm study. The focus is safety and tolerability (toxicity). Therefore, there are no results about factors and better or worse outcome. Population: In this study, Gross tumor volume is all known gross disease as demonstrated on end ventilation data set (30% phase as determined by Varian RPM or equivalent respiratory monitoring system) of the planning 4DCT using a lung window, and modified as deemed necessary based on PET/CT, diagnostic CT and other clinical studies.
  cubic centimeters | 42.9 [4.2 to 435.0]
iCTV (internal Clinical Target Volume) [Median (Full Range); unit: cubic centimeters] — This is phase I/II one arm study. The focus is safety and tolerability (toxicity). Therefore, there are no results about factors and better or worse outcome. Population: iCTV (internal Clinical Target Volume): Volume encompassing the Clinical Target Volume (CTV) and Internal Margin (IM). (iCTV = CTV + IM).
  In this study, the iCTV is envelope of motion of the CTV estimated by an 8-mm isotropic expansion of the iGTV to encompase microextensions of the tumor (iCTV = iGTV+8mm);
  cubic centimeters | 123 [14.3 to 786.6]
Pre-Treatment Pulmonary Function - FEV1 [Median (Full Range); unit: percentage of predicted (%)] — This is phase I/II one arm study. The focus is safety and tolerability (toxicity). Therefore, there are no results about factors and better or worse outcome. Population: There were 35 out of 38 patients treated under the protocol and evaluable for data analysis.
  percentage of predicted (%) | 48 [18 to 100]
Pre-Treatment Pulmonary Function - DLCO [Median (Full Range); unit: percentage of predicted (%)] — This is phase I/II one arm study. The focus is safety and tolerability (toxicity). Therefore, there are no results about factors and better or worse outcome. Population: There were 35 out of 38 patients treated under the protocol and evaluable for data analysis.
  percentage of predicted (%) | 49 [18 to 98]
Smoking History [Count of Participants; unit: Participants] — This is phase I/II one arm study. The focus is safety and tolerability (toxicity). Therefore, there are no results about factors and better or worse outcome. Population: There were 35 out of 38 patients treated under the protocol and evaluable for data analysis.
  Participants
    Yes | 31
    No | 4
Chronic Pulmonary Disease [Count of Participants; unit: Participants] — This is phase I/II one arm study. The focus is safety and tolerability (toxicity). Therefore, there are no results about factors and better or worse outcome. Population: There were 35 out of 38 patients treated under the protocol and evaluable for data analysis.
  Participants
    COPD | 16
    Emphysema | 3
    Pulmonary Fibrosis | 1
    Normal | 15
Tumor Histological Type [Count of Participants; unit: Participants] — This is phase I/II one arm study. The focus is safety and tolerability (toxicity). Therefore, there are no results about factors and better or worse outcome. Population: There were 35 out of 38 patients treated under the protocol and evaluable for data analysis.
  Participants
    Squamous cell carcinoma | 17
    Adenocarcinoma | 11
    Squamous cell carcinoma + adenocarcinoma | 1
    Neuroendocrine carcinoma | 1
    Non-small cell carcinoma | 5
Number of Participants with Tumor Location [Count of Participants; unit: Participants] — This is phase I/II one arm study. The focus is safety and tolerability (toxicity). Therefore, there are no results about factors and better or worse outcome. Population: There were 35 out of 38 patients treated under the protocol and evaluable for data analysis.
  Participants
    Central or Superior | 25
    Peripheral | 10
Number of Participants with Tumor size [Number; unit: participants] — This is phase I/II one arm study. The focus is safety and tolerability (toxicity). Therefore, there are no results about factors and better or worse outcome. Population: There were 35 out of 38 patients treated under the protocol and evaluable for data analysis.
  participants
    ≤3 cm | 13
    >3 cm ≤ 5 cm | 16
    >5 cm | 6
Number of Participants with Primary Tumor (T) Stage [Number; unit: participants] — This is phase I/II one arm study. The focus is safety and tolerability (toxicity). Therefore, there are no results about factors and better or worse outcome.
  American Joint Committee on Cancer (6th):
  T1:Tumor ≤3 cm in greatest dimension, T2:tumor>3 cm; involve: main bronchus, the visceral pleura or ≥ 2 cm to the Carina; atelectasis or pneumonia, T3:Invades: chest wall, diaphragm, mediastinal pleura, parietal pericardium, or tumor < 2 cm to the Carina, entire lung atelectasis or pneumonia, The earlier T staging, the better treatment outcome Population: There were 35 out of 38 patients treated under the protocol and evaluable for data analysis.
  participants
    T1:Tumor ≤3 cm in greatest dimension | 12
    T2:tumor>3 cm; involve: main bronchus, the viscera | 20
    T3 | 3
Number of Participants with Clinical Stage [Number; unit: participants] — AJCC (American Joint Committee on Cancer) TNM staging (6th): Stage IA :T1 N0 M0 Stage IB :T2 N0 M0 Stage IIA :T1 N1 M0 Stage IIB :T3 N0 M0. T describes size of tumor and any spread of cancer into nearby tissue; N describes spread of cancer to nearby lymph nodes; M describes metastasis (spread of cancer to other parts of body). Higher the T, N or M number, the larger the size of the tumor and/or more it has grown into nearby tissues, spread to lymph nodes or metastasized to distant organs, respectively. The earlier TNM staging, the better treatment outcome.
  participants
    IA | 12
    IB | 16
    IIA | 4
    IIB | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival and Progression Free Survival
Description: Chest CT with contrast (if possible) was used for evaluation of Local control. If is suspicious for recurrence by CT image, PET or PET/CT scan is required and biopsy is recommended to confirm the recurrence. Continuing CT or PET images follow up for un-confirmed recurrent disease. Timing of recurrence: at the time of first image (PET and/or CT) showing abnormalities. PET will use for progression free survival (PFS).
  Participants were followed up at 6 weeks after the completion of RT, every 3 months (±1 month) for 2 years, every 6 months (±1 month) for 3 years, and then annually. The Overall survival: time of registration to the last follow-up (f/u), or lost to f/u, or death. The PFS: time of registration to any local-regional recurrence or distant metastasis. Free local recurrence rate: time of registration to local recurrence. Free regional recurrence rate: time of registration to regional recurrence. Free distant metastasis rate: time of registration to distant metastasis.
Time Frame: The Overall survival (OS): time of registration to the last follow-up (f/u), or lost to f/u, or death up to 5 years. The progression free survival (PFS): time of registration to any local-regional recurrence or distant metastasis up to 5 years.
Population: Kaplan-Meier curves used for overall survival, progression-free survival, local recurrence-free survival, regional recurrence-free survival, and distant metastasis-free survival. Differences between pairs of Kaplan-Meier curves were using the log-rank test. The Fisher's exact test was used to compare local, regional, and distant recurrence rates.
Measure: Number; unit: percentage of participants (%)
Arm/Group | Dose-escalated Proton Therapy for Early-stage Non-small Cell l
Number analyzed (Participants) | 35
percentage of participants (%)
  Overall Survival rate : 1 year | 85.70
  Overall Survival rate : 2 year | 60
  Overall Survival rate : 3 year | 42.90
  Overall Survival rate : 5 year | 28.10
  Progression Free Survival rate : 1 year | 80
  Progression Free Survival rate : 2 year | 64.40
  Progression Free Survival rate : 3 year | 53.60
  Progression Free Survival rate : 5 year | 53.60
  free local recurrence rate 5-year | 85
  free from regional recurrence rate: 5-year | 89.20
  free from distant metastasis rate: 5-year | 56

ADVERSE EVENTS:
Time Frame: From the time of registration to the time of the adverse event start date, up to 5 years.
Description: Grade > 3 acute and chronic toxicities by Common Terminology Criteria for Adverse Events, version 3.0 (CTCAE 3.0) will be analyzed.
Arm/Group | Dose-escalated Proton Therapy for Early-stage Non-small Cell l
All-Cause Mortality (participants affected / at risk) | 30/35
Serious Adverse Events (participants affected / at risk) | 2/35
Other Adverse Events (participants affected / at risk) | 0/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose-escalated Proton Therapy for Early-stage Non-small Cell l (N=35)
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Esophagitis (Gastrointestinal disorders) | 0
Atrial fibrillation (Cardiac disorders) | 0
Rib fracture (Musculoskeletal and connective tissue disorders) | 0
Chest wall pain (General disorders) | 0

LIMITATIONS AND CAVEATS:
This is phase I/II one arm study. The focus is safety and tolerability (toxicity). Therefore, there are no results about factors and better or worse outcome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2010-04-19): https://cdn.clinicaltrials.gov/large-docs/40/NCT00495040/Prot_SAP_000.pdf